CLINICAL TRIAL: NCT05050292
Title: Cognitive Stimulation Intervention Program for Insomniacs and Its Benefit on Sleep Quality, Executive Functions and Quality of Life
Brief Title: Cognitive Stimulation and Sleep Quality. An Innovative Intervention for Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Antonio de Nebrija (Other)
Collaborators: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Jon Andoni Duñabeitia, Director, Universidad Antonio de Nebrija
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBEF21
Record Dates: First submitted 2021-09-06; First posted 2021-09-20 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Insomnia; Insomnia Type; Sleep Disorder
Keywords: Insomnia; Cognitive stimulation; Cognitive intervention; Sleep disorder; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: The intervention will be carried out through the CogniFit® online platform so participants will access it from home using a personal computer or smart device. The training will last for a total of 8 weeks (40 training sessions), with five consecutive training days per week (Monday to Friday). Since this process is autonomous, participants will be contacted periodically (a minimum of one phone call per week) to ensure adherence and check that they have not had any incidence. The platform will records participants' performance, providing researchers with real-time feedback on the performance of each participant.
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly assigned to one out of two groups (control/experimental).
  The activities presented to Group 1 (experimental group) will target executive functions skills and will be automatically adjusted in difficulty and requirement according to each participant's performance so that a maximum cognitive effort is always required.
  The activities for Group 2 (active control group) will be of constant difficulty throughout the intervention and will not target the intended cognitive processes (namely, they will target orthogonal unrelated aspects).
  Participants and researchers are blind to whether they are in the intervention or the control group. In this way, placebo or waiting-list effects are avoided.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Activities are designed to target specific cognitive skills (attention, perception, inhibition).
  An internal algorithm of the cognitive stimulation platform will adjust the activities' difficulty depending on the participant's performance, always demanding a maximum cognitive effort.
  Interventions: Other: Personalized cognitive stimulation
- Control Group (Active Comparator): Painting and artistic activities not designed to target specific cognitive skills.
  The internal algorithm will be deactivated, so the cognitive stimulation activities will be of constant difficulty throughout the intervention.
  Interventions: Other: Sham cognitive stimulation

INTERVENTIONS:
Other: Personalized cognitive stimulation — Online gamified activities designed to stimulate cognitive functions (specifically executive function) will be carried out through a mobile application or web browser.
  Performance feedback will be shown after each activity.
  Other Names: CogniFit's personalized brain training
  Arms: Experimental Group
Other: Sham cognitive stimulation — Non-therapeutic online games based on artistic and creative tasks. Activities will match in duration to those of the experimental intervention.
  Performance feedback will be shown after each game.
  Arms: Control Group

SUMMARY:
The purposes of this study are a) to investigate the effect of a personalized and computerized cognitive stimulation program on sleep quality, cognitive performance, and quality of life; and b) verify if cognitive stimulation can be used as a non-pharmacological alternative to improve the quality of sleep in individuals who have insomnia.

DETAILED DESCRIPTION:
Phase I/II was designed to determine the safety of the training, the maximum tolerated training time per session, and the needed training sessions to obtain significant cognitive performance improvement prior to beginning with the cognitive stimulation intervention program (Phase III).

Phase I/II

Through a 3+3 design, a dose-escalation trial will be set. Participants will be tested across subsequent training blocks of 15 minutes each, reporting experienced fatigue or adverse effects after every block. The safe training dose will be set to a block before extreme fatigue or a notable adverse effect has been reported by two or more participants.

Once a safety training time has been established, 20 participants will engage in a 15-day training effectiveness assessment. An evaluation day and a training day will be interspersed so that participants will complete a total of 7 training sessions (days 2, 4, 6, 8, 10, 12, and 14) and 8 evaluation sessions (days 1, 3, 5, 7, 9, 11, 13, and 15).

A psychologist will be supervising every step of the process at all times.

Phase III

A total of 120 persons with insomnia will undergo an 8-week cognitive stimulation program, five consecutive days per week. Eligible participants will be randomized in a 1:1 ratio to an intervention or control group. Activities duration per day will be as set on phase I.

This final phase is set to be an online home-based stage, although the responsible psychologist will periodically contact participants via telephone.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed by Insomnia Disorder [307.42 (F51.01)]:

A. A predominant complaint of dissatisfaction with sleep quantity or quality, associated with one (or more) of the following symptoms:

1. Difficulty initiating sleep. (In children, this may manifest as difficulty initiating sleep without caregiver intervention.)
2. Difficulty maintaining sleep, characterized by frequent awakenings or problems returning to sleep after awakenings. (In children, this may manifest as difficulty returning to sleep without caregiver intervention.)
3. Early-morning awakening with inability to return to sleep.

B. The sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning.

C. The sleep difficulty occurs at least 3 nights per week.

D. The sleep difficulty is present for at least 3 months.

E. The sleep difficulty occurs despite adequate opportunity for sleep.

F. The insomnia is not better explained by and does not occur exclusively during the course of another sleep-wake disorder (e.g., narcolepsy, a breathing-related sleep disorder, a circadian rhythm sleep-wake disorder, a parasomnia).

G. The insomnia is not attributable to the physiological effects of a substance (e.g., a drug of abuse, a medication).

H. Coexisting mental disorders and medical conditions do not adequately explain the predominant complaint of insomnia.

Exclusion Criteria:

* Have another sleep-wake disorder (e.g., narcolepsy, restless leg syndrome, a breathing-related sleep disorder, a circadian sleep-wake rhythm disorder, a parasomnia).
* Presence of a relevant medical, psychiatric or neurological disorder.
* Significant visual or motor impairments.
* History of alcohol or drug abuse or dependence.
* Caffeine consumption (more than 150mg per day, that is, approximately 3 cups of espresso or a cup of American coffee).
* Alcohol consumption (more than 250ml per day, that is, around a pint of beer, a glass of wine, or a shot of liquor).
* Use of medications with stimulant action, except sedatives or hypnotics prescribed for sleep.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-03-16 (Estimated); Study Completion 2023-03-16 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Sleep quality on the Pittsburgh Sleep Quality Index at Week 8 | 1 day before starting the intervention and 1 day after finishing the intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality. Change = (Week 8 Score - Baseline Score).
Change from Baseline in Insomnia on the Insomnia Severity Index at Week 8 | 1 day before starting the intervention and 1 day after finishing the intervention
  The Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. It comprises seven items assessing the perceived severity of difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Possible scores ranges from 0 (No clinically significant insomnia) to 28 (Clinically insomnia - Severe). Change = (Week 8 Score - Baseline Score).
Change from Baseline in Quality of life on Measuring Quality of Life | The World Health Organization - abridged version | 1 day before starting the intervention and 1 day after finishing the intervention
  The Measuring Quality of Life | The World Health Organization - abridged version (WHOQOL-BREF) is a generic questionnaire to measure the quality of life created by the Study Group on Quality of Life of the World Health Organization. It has 26 questions, two general questions on the quality of life and satisfaction with the state health, and 24 questions grouped into four areas or domains: Physical Health, Psychological Health, Social Relations and Environment. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval. Possible scores for each domain ranges from 0 (poor perceived quality of life) to 100 (greater perceived quality of life). Change = (Week 8 Score - Baseline Score).

SECONDARY OUTCOMES:
Change from Baseline in Executive function on Behavior Rating Inventory of Executive Function-Adult Version at Week 8 | 1 day before starting the intervention and 1 day after finishing the intervention
  The Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) is a standardised measure that captures views of an adult's executive functions or self-regulation in his or her everyday environment. Only the self-report format will be used. The BRIEF-A is composed of 75 items within nine theoretically and empirically derived clinical scales that measure various aspects of executive functioning; Inhibit, Self-Monitor, Plan/Organise, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, Organisation of Materials. The clinical scales form two broader indexes: Behavioral Regulation (BRI) and Metacognition (MI), and these indexes form the overall summary score, the Global Executive Composite (GEC). Also includes three validity scales (Negativity, Inconsistency, and Infrequency). It takes approximately 10-15 minutes to administer. All 75 items are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). Raw scores for each scale are summed
Change from Baseline in Depressive symptoms on The Beck Depression Inventory-II at Week 8 | 1 day before starting the intervention and 1 day after finishing the intervention
  The Beck Depression Inventory-II (BDI-II) is a 21-item, self-report inventory designed to measure the frequency and severity of depressive symptoms. Items include somatic-affective symptoms as well as cognitive symptoms. Possible scores ranges from 0 (no depressive symptoms) to 63 (severe depression). Change = (Week 8 Score - Baseline Score).
Change from Baseline in Anxiety symptoms on the State-Trait Anxiety Inventory at Week 8 | 1 day before starting the intervention and 1 day after finishing the intervention
  The State-Trait Anxiety Inventory (STAI) is a self-report that assesses two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Only the 20 items referred to state anxiety will be administered. Possible scores ranges from 0 (no anxiety) to 60 (severe anxiety). Change = (Week 8 Score - Baseline Score).
Change from Baseline in worrying on The Penn State Worry Questionnaire at Week 8 | 1 day before starting the intervention and 1 day after finishing the intervention
  The Penn State Worry Questionnaire (PSWQ) is a 16-item questionnaire that aims to measure the trait of worry. The items on the scale assess the occurrence, intrusiveness, pervasiveness, and other characterizing features of an individual's experience with worry. The scale has been shown to identify worry, over and above anxiety and depression. Items are rated on a five-point scale: 1-Not at all typical of me to 5-Very typical of me. Possible scores ranges from 16 (low worry) to 80 (high worry). Change = (Week 8 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Overall Officials: Jon A Duñabeitia, Study Director — Universidad Nebrija; Jose L Tapia, Principal Investigator — Univerisdad Nebrija
Locations (1):
- Hospital Universitario de la Ribera, Alzira, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Due to the institutional restrictions that regulate the data protection of patients in the Spanish public health system, it is not possible for the investigators to share any individual participant data.

REFERENCES:
- [Background] Bastien CH, St-Jean G, Morin CM, Turcotte I, Carrier J. Chronic psychophysiological insomnia: hyperarousal and/or inhibition deficits? An ERPs investigation. Sleep. 2008 Jun;31(6):887-98. doi: 10.1093/sleep/31.6.887. PMID 18548835
- [Background] Bastien CH, Vallieres A, Morin CM. Precipitating factors of insomnia. Behav Sleep Med. 2004;2(1):50-62. doi: 10.1207/s15402010bsm0201_5. PMID 15600224
- [Background] Corsi-Cabrera M, Figueredo-Rodriguez P, del Rio-Portilla Y, Sanchez-Romero J, Galan L, Bosch-Bayard J. Enhanced frontoparietal synchronized activation during the wake-sleep transition in patients with primary insomnia. Sleep. 2012 Apr 1;35(4):501-11. doi: 10.5665/sleep.1734. PMID 22467988
- [Background] Espie CA. Insomnia: conceptual issues in the development, persistence, and treatment of sleep disorder in adults. Annu Rev Psychol. 2002;53:215-43. doi: 10.1146/annurev.psych.53.100901.135243. PMID 11752485
- [Background] Haimov I, Shatil E. Cognitive training improves sleep quality and cognitive function among older adults with insomnia. PLoS One. 2013;8(4):e61390. doi: 10.1371/journal.pone.0061390. Epub 2013 Apr 5. PMID 23577218
- [Background] Harvey AG. A cognitive model of insomnia. Behav Res Ther. 2002 Aug;40(8):869-93. doi: 10.1016/s0005-7967(01)00061-4. PMID 12186352
- [Background] Harvey AG, Tang NK. (Mis)perception of sleep in insomnia: a puzzle and a resolution. Psychol Bull. 2012 Jan;138(1):77-101. doi: 10.1037/a0025730. Epub 2011 Oct 3. PMID 21967449
- [Background] Aasvik J, Stiles TC, Woodhouse A, Borchgrevink P, Inge Landro N. The Effect of Insomnia on Neuropsychological Functioning in Patients with Comorbid Symptoms of Pain, Fatigue, and Mood Disorders. Arch Clin Neuropsychol. 2018 Feb 1;33(1):14-23. doi: 10.1093/arclin/acx040. PMID 28453603
- [Background] Fortier-Brochu E, Morin CM. Cognitive impairment in individuals with insomnia: clinical significance and correlates. Sleep. 2014 Nov 1;37(11):1787-98. doi: 10.5665/sleep.4172. PMID 25364074
- [Background] Brownlow JA, Miller KE, Gehrman PR. Insomnia and Cognitive Performance. Sleep Med Clin. 2020 Mar;15(1):71-76. doi: 10.1016/j.jsmc.2019.10.002. Epub 2019 Nov 27. PMID 32005351
- [Background] Leerssen J, Wassing R, Ramautar JR, Stoffers D, Lakbila-Kamal O, Perrier J, Bruijel J, Foster-Dingley JC, Aghajani M, van Someren EJW. Increased hippocampal-prefrontal functional connectivity in insomnia. Neurobiol Learn Mem. 2019 Apr;160:144-150. doi: 10.1016/j.nlm.2018.02.006. Epub 2018 Feb 12. PMID 29448003
- [Background] Perlis ML, Giles DE, Mendelson WB, Bootzin RR, Wyatt JK. Psychophysiological insomnia: the behavioural model and a neurocognitive perspective. J Sleep Res. 1997 Sep;6(3):179-88. doi: 10.1046/j.1365-2869.1997.00045.x. PMID 9358396
- [Background] Riemann D, Nissen C, Palagini L, Otte A, Perlis ML, Spiegelhalder K. The neurobiology, investigation, and treatment of chronic insomnia. Lancet Neurol. 2015 May;14(5):547-58. doi: 10.1016/S1474-4422(15)00021-6. Epub 2015 Apr 12. PMID 25895933
- [Background] Thomas M, Sing H, Belenky G, Holcomb H, Mayberg H, Dannals R, Wagner H, Thorne D, Popp K, Rowland L, Welsh A, Balwinski S, Redmond D. Neural basis of alertness and cognitive performance impairments during sleepiness. I. Effects of 24 h of sleep deprivation on waking human regional brain activity. J Sleep Res. 2000 Dec;9(4):335-52. doi: 10.1046/j.1365-2869.2000.00225.x. PMID 11123521
- [Derived] Tapia JL, Puertas FJ, Dunabeitia JA. Digital Therapeutics for Insomnia: Assessing the Effectiveness of a Computerized Home-Based Cognitive Stimulation Program. J Integr Neurosci. 2023 Feb 14;22(2):34. doi: 10.31083/j.jin2202034. PMID 36992590
- [Derived] Tapia JL, Puertas FJ, Dunabeitia JA. Study Protocol for a Randomized Controlled Trial Assessing the Effectiveness of Personalized Computerized Cognitive Training for Individuals With Insomnia. Front Behav Neurosci. 2022 Feb 28;16:779990. doi: 10.3389/fnbeh.2022.779990. eCollection 2022. PMID 35296055